CLINICAL TRIAL: NCT04941768
Title: Real-world Evaluation of Efficacy and Safety With Avelumab (BAVENCIO®) + Axitinib (INLYTA®) in Patients With aRCC in Multiple EU Countries (AVION)
Brief Title: An Observational Study to Evaluate the Efficacy and Safety of Avelumab + Axitinib Combination in Participants With aRCC (AVION)
Status: Completed | Type: Observational
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Healthcare Germany GmbH, an affiliate of Merck KGaA, Darmstadt, Germany (Unknown)
Responsible Party: Sponsor
Other Study IDs: MS100070_0110
Record Dates: First submitted 2021-06-23; First posted 2021-06-28 (Actual); Results first posted 2025-11-28 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Renal Cell
Keywords: Axitinib; Renal cell carcinoma; Avelumab; BAVENCIO®; INLYTA®
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Avelumab + Axitinib: There will not be any study-specific interventions in this study. Participants with advanced RCC receiving 800 milligrams (mg) of Avelumab intravenously every 2 weeks in combination with 5 mg of Axitinib orally twice per day in accordance with the terms of marketing authorization for the first-line therapy as per the current clinical practice will be observed for 24 months in this study.

SUMMARY:
The main purpose of this study is to expand knowledge on the effectiveness of Avelumab intravenous infusion in combination with Axitinib as the first-line therapy in participants with advanced renal-cell carcinoma (aRCC) in addition to the safety and tolerability under routine conditions of daily clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Participants with the Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Participants with a histologically confirmed diagnosis of RCC with any histological origin
* Participants with a locally advanced/metastatic disease (that is [ie], newly diagnosed Stage 4 RCC per American Joint Committee on Cancer) or has recurrent disease
* Participants has received 1 or 2 cycles of Avelumab plus Axitinib treatment as a first-line therapy according to the approved Summary of Product Characteristics (SmPC)
* Participants willing to sign the written informed consent form (ICF) to participate in this study

Exclusion Criteria:

* Participants with contraindications for Avelumab or Axitinib according to the approved SmPC
* Participants who have participated in any interventional clinical study of a drug or device within 28 days prior to the start of Avelumab plus Axitinib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with a confirmed diagnosis of advanced RCC will be observed in this study.
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2021-08-09 (Actual); Primary Completion 2024-08-08 (Actual); Study Completion 2025-04-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (61):
- Belgium (3):
  - Imelda Ziekenhuis, Bonheiden
  - AZ KLINA, Brasschaat
  - AZ Sint-Jan, Bruges
- Germany (40):
  - Klinikum St. Marien Amberg, Amberg
  - Klinikum Aschaffenburg Medizinische Klinik, Aschaffenburg
  - Zentrum für urologische Onkologie, Berlin
  - Biberach, Biberach an der Riss
  - Evangelisches Klinikum Bethel, Bielefeld
  - Evangelisches Krankenhaus Bielefeld, Bielefeld
  - Urologie im Schlosscarree, Braunschweig
  - Donauisar Klinikum Deggendorf, Deggendorf
  - Urologische Gemeinschaftspraxis, Dresden
  - St. Georg Klinikum Eisenach gGmbH, Eisenach
  - Universitatsklinikum Erlangen, Erlangen
  - Universitaetsklinikum Essen Uroonkologie, Essen
  - Klinikum Friedrichshafen GmbH daVinci® -Zentrum Bodensee, Friedrichshafen
  - Onkologische GP Dres. Wilke/Wagner/Petzoldt, Fürth
  - Onkologische SP Praxis Fürth, Fürth
  - MVZ Onkologische Kooperation Harz GbR, Goslar
  - Praxis Dr. Maas, Halberstadt
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Medizinische Hochschule Hannover, Hanover
  - Vinzenzkrankenhaus Hannover, Hanover
  - Praxis Kretz, Heinsberg
  - Universitätskinderklinik Jena, Jena
  - Urologische Praxis Dr. Ralf Eckert, L.-Eisleben
  - Urologische Praxis Dipl.-Med. Susanne Kloß, Luckenwalde
  - Universitatsklinik Schleswig-Holstein, Lübeck
  - Schwerpunktpraxis für Hämatologie und Onkologie, Magdeburg
  - Johannes Wesling Klinikum Minden der Mühlenkreiskliniken (AöR), Minden
  - Uniklinikum Münster, Münster
  - University of Munster, Münster
  - Klinikum Osnabrück GmbH, Osnabrück
  - Marienhospital Osnabrück - Standort Natruper Holz, Osnabrück
  - Paracelsus Klinik Osnabrück, Osnabrück
  - medius Klinik Ostfildern-Ruit, Ostfildren
  - Wissenschaftskontor Nord GmbH & Co. KG, Rostock
  - GPR Klinikum Rüsselsheimg GmbH, Rüsselsheim am Main
  - SRH Kliniken Landkreis Sigmaringen (DEU), Sigmaringen
  - Hämatologie und Onkologie Stolberg, Stolberg
  - Praxis Troisdorf, Troisdorf
  - Medizinische Studiengesellschaft Nord-West GmbH, Westerstede
  - Lahn Dill Kliniken GmbH, Wetzlar
- Greece (17):
  - Gen. Hos. "Alexandra", Athens
  - General Hospital of Athens G.Gennimatas, Athens
  - Henry Dunant Hospital Center, Athens
  - University Hospital of Athens Sotiria, Athens
  - Attikon Hospital, Attiki
  - Attikon, Chaïdári
  - General Hospital "Venizelio", Heraklion
  - University Hospital of Ioannina, Ioannina
  - Kavala General Hospital, Kavala
  - University Hospital of Larissa, Larissa
  - General Hospital of Patras "o Agios Andreas", Pátrai
  - Metaxa Hospital, Piraeus
  - Metropolitan Hospital Greece, Piraeus
  - Agios Loukas Hospital, Thessaloniki
  - Bioclinic (GRC), Thessaloniki
  - Papageorgiou Hospital, Thessaloniki
  - Saint Luke Hospital, Thessaloniki
- Regional Oncology Dispensary - Irkutsk, Irkutsk, Russia

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS100070_0110
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The results reported are based on the primary analyses at the 12-months cut-off.
Groups:
- Avelumab + Axitinib: Participants with advanced renal cell carcinoma (RCC) received 800 milligrams (mg) of Avelumab intravenously every 2 weeks (Q2W) in combination with 5 mg of Axitinib orally twice per day in accordance with the terms of marketing authorization for the first-line therapy as per the current clinical practice were observed for 24 months in this study.
Period: Overall Study
Arm/Group | Avelumab + Axitinib
Started | 105
Completed | 18
Not Completed | 87
Not completed — Lost to Follow-up | 10
Not completed — Death | 24
Not completed — Progressive Disease | 4
Not completed — Withdrawal by Subject | 4
Not completed — Other | 3
Not completed — Treatment ongoing | 21
Not completed — Off treatment and in follow-up | 21

BASELINE CHARACTERISTICS:
Population: Analysis set (AS) included all eligible participants who provided written informed consent and received 1 or 2 cycles of avelumab plus axitinib treatment as a first-line therapy prior to informed consent.
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 104
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 73
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 104

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS) Rate
Description: OS rate was defined as the percentage of participants who are alive at 12 months after the index date. Percentage of participants alive at the time of outcome assessment (12 months) were calculated as per the Kaplan-Meier (KM) approach. The index date (baseline visit) was defined as the date of first administration after obtaining informed consent of avelumab plus axitinib therapy to participants with advanced RCC.
Time Frame: At 12 months after index date (baseline visit as reported in the electronic case report form [eCRF])
Population: AS included all eligible participants who provided written informed consent and received 1 or 2 cycles of avelumab plus axitinib treatment as a first-line therapy prior to informed consent.
Measure: Number; unit: Percentage of Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 104
Percentage of Participants | 82.7

2. Secondary Outcome: OS Rate
Time Frame: At 24 months after index date (baseline visit as reported in the eCRF)
Reporting Status: Not Posted, anticipated posting 2026-04

3. Secondary Outcome: Duration of OS
Time Frame: At 24 months after index date
Reporting Status: Not Posted, anticipated posting 2026-04

4. Secondary Outcome: Objective Response Rate (ORR) Assessed by Investigator up to 24 Months After the Index Date
Time Frame: up to 24 months after the index date
Reporting Status: Not Posted, anticipated posting 2026-04

5. Secondary Outcome: Disease Control Rate (DCR) Assessed by Investigator up to 24 Months After the Index Date
Time Frame: up to 24 months after the index date
Reporting Status: Not Posted, anticipated posting 2026-04

6. Secondary Outcome: Duration of Response (DoR) According to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1
Time Frame: up to 24 months after the index date
Reporting Status: Not Posted, anticipated posting 2026-04

7. Secondary Outcome: Progression-free Survival (PFS) According to Response Evaluation Criteria in Solid Tumours (RECIST) Version 1.1 Assessed by Investigator
Description: PFS time was defined as the time from index date to the date of the first documentation of objective progressive disease (PD) or death due to any cause, whichever occurred first. Per RECIST version 1.1, PD was defined as at least a 20 percent (%) increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 millimeter (mm). The appearance of one or more new lesions was also considered PD. The tumor response was determined according to RECIST version 1.1 and assessed by the investigator. PFS was calculated based on KM method. The index date (baseline visit) was defined as the date of first administration after obtaining informed consent of avelumab plus axitinib therapy to participants with advanced RCC.
Time Frame: From the index date to the date of disease progression or death from any cause, whichever occurred first (assessed up to 12 months after index date)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 104
months | 11.3 [8.1 to NA] — Here "NA" means the upper limit of 95% confidence interval could not be estimated due to small number of death events resulting large variability and therefore the upper 95% confidence limits of KM survival estimate remaining above 50%.

8. Secondary Outcome: Progression-free Survival 2 (PFS2) According to RECIST Version 1.1 Assessed by Investigator
Description: PFS2 was defined as time interval from the index date to the date of disease progression on second-line treatment or death from any cause, whichever occurred first. Per RECIST version 1.1, PD was defined as at least a 20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions was also considered PD. The tumor response will be determined according to RECIST version 1.1 and assessed by the investigator. PFS2 was calculated based on Kaplan Meier method. The index date (baseline visit) was defined as the date of first administration after obtaining informed consent of avelumab plus axitinib therapy to participants with advanced RCC.
Time Frame: From the index date to the date of disease progression on second-line treatment or death from any cause, whichever occurred first (assessed up to 12 months after index date)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 104
months | NA [11.8 to NA] — Here "NA" means median and upper limit of 95% confidence interval could not be estimated due to small number of death events resulting large variability and therefore the upper 95% confidence limits of KM survival estimate remaining above 50%.

9. Secondary Outcome: Change From Baseline in National Comprehensive Cancer Network/Functional Assessment of Cancer Therapy-Kidney Symptom Index 19 (NCCN-FACT FKSI-19) Total Score
Description: NCCN-FACT FKSI-19, a validated, disease-specific questionnaire for RCC. It includes 19 items across four domains,Disease-Related Symptoms-Physical (DRS-P), Disease-Related Symptoms-Emotional (DRS-E), Treatment Side Effects (TSE), and Functional Wellbeing (FWB), based on symptoms experienced over past 7 days. Responses were recorded on 5-point Likert scale (0 = not at all to 4 = very much), yielding a total score from 0 to 76, higher scores reflecting better quality of life. A negative mean change in score indicated worsening condition. Domain score ranges and directionality: DRS-P: 0-48, higher scores = fewer physical symptoms; DRS-E: 0-4, higher = fewer emotional symptoms; TSE: 0-32, higher = more severe side effects; FWB: 0-12, higher = better functional wellbeing. As per NCCN-FACT FKSI-19 scoring guidelines, the total Health-related quality of life (HRQoL) score (range 0-76) was calculated as sum of single items scores multiplied by 19 and divided by the number of items completed.
Time Frame: Index date (Baseline), at 6, 12, 18, 24, 30, 36, 42, 48, 54, 60, 66, 72, 78, 84, 90 and 96 weeks
Population: AS included all eligible participants who provided written informed consent and received 1 or 2 cycles of avelumab plus axitinib treatment as a first-line therapy prior to informed consent. Here" overall number of participants analyzed signified" participants who were evaluable for this outcome measure and "number analyzed" signifies participants who were evaluable at specified timepoints.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 95
scores on a scale
  Baseline | 58.3 (9.64)
  6 Weeks: number analyzed (Participants) | 76
  6 Weeks | -0.2 (8.38)
  12 Weeks: number analyzed (Participants) | 71
  12 Weeks | -1.1 (10.36)
  18 Weeks: number analyzed (Participants) | 63
  18 Weeks | -0.6 (9.42)
  24 Weeks: number analyzed (Participants) | 60
  24 Weeks | -0.3 (10.04)
  30 Weeks: number analyzed (Participants) | 51
  30 Weeks | -1.4 (10.08)
  36 Weeks: number analyzed (Participants) | 49
  36 Weeks | -0.4 (7.89)
  42 Weeks: number analyzed (Participants) | 44
  42 Weeks | -0.8 (8.58)
  48 Weeks: number analyzed (Participants) | 44
  48 Weeks | -0.8 (10.06)
  54 Weeks: number analyzed (Participants) | 42
  54 Weeks | -0.7 (10.29)
  60 Weeks: number analyzed (Participants) | 39
  60 Weeks | -0.4 (10.47)
  66 Weeks: number analyzed (Participants) | 30
  66 Weeks | -0.6 (11.21)
  72 Weeks: number analyzed (Participants) | 25
  72 Weeks | -1.1 (8.94)
  78 Weeks: number analyzed (Participants) | 27
  78 Weeks | -1.3 (8.86)
  84 Weeks: number analyzed (Participants) | 24
  84 Weeks | -1.0 (9.87)
  90 Weeks: number analyzed (Participants) | 16
  90 Weeks | -1.3 (9.67)
  96 Weeks: number analyzed (Participants) | 13
  96 Weeks | 1.4 (9.42)

10. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs), Serious TEAEs, Related TEAEs, TEAEs Leading to Permanent Treatment Discontinuation and TEAEs Leading to Death According to Medical Dictionary for Regulatory Activities (MedDRA)
Time Frame: From the index date up to 90 days post discontinuation of avelumab plus axitinib or completion of the 24 months (i.e., end of the study) follow-up from the index date, whichever occured first
Reporting Status: Not Posted

11. Secondary Outcome: Number of Participants With Adverse Events (AEs) Based on Severity According to National Cancer Institute - Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
Time Frame: as for outcome 10
Reporting Status: Not Posted, anticipated posting 2026-04

12. Secondary Outcome: Time to Therapy Discontinuation Due to AE Greater Than or Equal to (>=) Grade-3
Time Frame: From index date up to Month 24
Reporting Status: Not Posted, anticipated posting 2026-04

13. Secondary Outcome: Duration of Avelumab Plus Axitinib Therapy Among Participants Who Discontinued the Study Drugs Due to All-Cause AEs >= Grade 3
Time Frame: Time from first dose of study drug up to Month 24
Reporting Status: Not Posted, anticipated posting 2026-04

14. Secondary Outcome: Time to Onset of All-cause AEs
Time Frame: From index date up to Month 24
Reporting Status: Not Posted, anticipated posting 2026-04

15. Secondary Outcome: Duration of All-cause AEs
Time Frame: From index date up to Month 24
Reporting Status: Not Posted, anticipated posting 2026-04

16. Secondary Outcome: Percentage of Participants With Therapy Modifications Due to Adverse Event Related to Avelumab Plus Axitinib Therapy
Time Frame: From index date up to Month 24
Reporting Status: Not Posted, anticipated posting 2026-04

17. Secondary Outcome: Number of Participants With Different Types of Medical Intervention or Medications Used for the Management of TEAEs Related to Avelumab Plus Axitinib Therapy
Description: Number of participants with different types of medical intervention or medications used for the management of TEAE related to avelumab plus axitinib therapy (e.g., use of corticosteroids, antihypertensive therapy, treatment for thyroid dysfunction, measures to decrease hemoglobin, and hematocrit) was reported.
Time Frame: From index date upto 12 months after the index date
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 104
Participants
  Any related TEAE managed with concomitant medications | 47
  Any related TEAE managed with concomitant procedures | 6
  Any related TEAE managed with corticosteroids, immunosuppressants, or hormonal therapy | 11

18. Secondary Outcome: Percentage of Participants Receiving Later-line Therapy
Time Frame: From index date up to Month 24
Reporting Status: Not Posted, anticipated posting 2026-04

19. Secondary Outcome: Time to Second-line Therapy Initiation
Description: Time to 2nd line treatment was calculated as: (2nd line treatment start date - last dose of Avelumab plus Axitinib + 1)/30.4375.
Time Frame: Time from Avelumab plus Axitinib therapy discontinuation to the initiation of second-line therapy, up to Month 12
Population: AS included all eligible participants who provided written informed consent and received 1 or 2 cycles of avelumab plus axitinib treatment as a first-line therapy prior to informed consent. Here" overall number of participants analyzed signified" participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Avelumab + Axitinib
Number analyzed (Participants) | 12
months | 0.3 (0.40)

20. Secondary Outcome: Number of Participants With Patient-reported Potential Signs and Symptoms of Immune-related AEs
Time Frame: From index date up to Month 24
Reporting Status: Not Posted, anticipated posting 2026-04

ADVERSE EVENTS:
Time Frame: From index date up to 12 months after the index date
Description: AS included all eligible participants who provided written informed consent and received 1 or 2 cycles of avelumab plus axitinib treatment as a first-line therapy prior to informed consent and All-Cause Mortality data was assessed in all enrolled participants.
Arm/Group | Avelumab + Axitinib
All-Cause Mortality (participants affected / at risk) | 24/105
Serious Adverse Events (participants affected / at risk) | 38/104
Other Adverse Events (participants affected / at risk) | 80/104
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Axitinib (N=104)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
COVID-19 (Infections and infestations) | 2
Gallbladder abscess (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Diarrhoea 3 ( 2.9) (Gastrointestinal disorders) | 3
Diverticular perforation (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Post procedural infection (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Disease progression (General disorders) | 1
Gait disturbance (General disorders) | 1
Hypothermia (General disorders) | 1
Pain (General disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myositis (Musculoskeletal and connective tissue disorders) | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 1
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 1
Haemorrhage intracranial (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Monoparesis (Nervous system disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Myocarditis (Cardiac disorders) | 1
Autoimmune hepatitis (Hepatobiliary disorders) | 1
Cholecystitis acute (Hepatobiliary disorders) | 1
Immune-mediated hepatitis (Hepatobiliary disorders) | 1
Blood creatinine increased (Investigations) | 2
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1
Acute kidney injury (Renal and urinary disorders) | 2
End stage renal disease (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 2
Hypertensive crisis (Vascular disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Cataract (Eye disorders) | 1
Hypersensitivity (Immune system disorders) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Ureteral stent insertion (Surgical and medical procedures) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Cardiac failure chronic (Cardiac disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Avelumab + Axitinib (N=104)
Diarrhoea (Gastrointestinal disorders) | 26
Nausea (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 7
Fatigue (General disorders) | 17
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9
Back pain (Musculoskeletal and connective tissue disorders) | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 9
Pruritus (Skin and subcutaneous tissue disorders) | 8
Weight decreased (Investigations) | 6
Hypertension (Vascular disorders) | 11
Hypothyroidism (Endocrine disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2023-04-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04941768/Prot_000.pdf
  • Statistical Analysis Plan (2021-11-24): https://cdn.clinicaltrials.gov/large-docs/68/NCT04941768/SAP_001.pdf